CLINICAL TRIAL: NCT06510920
Title: Effects of Aerobic Exercise on Executive Function Among Obese Children
Brief Title: The Purpose of This Research is to Investigate the Effects of Aerobic Exercise on Executive Function in Obese Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jing Xin (Other)
Responsible Party: Sponsor-Investigator, Jing Xin, PHD, Universiti Putra Malaysia
Organization: Universiti Putra Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: - JKEUPM-2024-232
Record Dates: First submitted 2024-06-27; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Executive Function Disorder; Obesity, Childhood
Keywords: Executive function; Obese Children; Aerobic Exercise; Mental health
MeSH Terms: conditions — Pediatric Obesity; Psychological Well-Being | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese children aerobic exercise intervention group (Experimental): Aerobic exercise intervention on children obesity in the experimental group, the form of aerobic exercise for football and volleyball training, strength control in moderate intensity, time 1 hour, twice a week.
  Interventions: Behavioral: Aerobic exercise
- Obese children of control group (No Intervention): Control group in obese children will be conducted in normal school physical education, in addition to no other exercise intervention.

INTERVENTIONS:
Behavioral: Aerobic exercise — The mixed design scheme of football and volleyball sports technology and competition will be adopted.aerobic exercise intensity will be moderate-intensity aerobic exercise load , and the intervention time was 12 weeks, 60 minutes each time, twice a week. The main preparation activities were jogging and special preparation activities (10 minutes), and the main part was technical teaching combined with competition (60 minutes).The end part is mostly jogging and stretching (10 minutes). Two subjects in each group were selected to wear Decathlon Bluetooth heart rate band, and the exercise intensity was controlled by detecting the heart rate of the subjects.
  Arms: Obese children aerobic exercise intervention group

SUMMARY:
The goal of this clinical trial is to learn if aerobic exercise improves executive functioning in obese children. It will also understand the effects of aerobic exercise on executive functioning in obese children. The main questions it aims to answer are:

1. What are the levels of executive functioning(inhibitory function, working memory, and cognitive flexibility) in normal-weight and obese children aged 8-10 years?
2. What are the differences on executive function before and after aerobic exercise intervention among obese children?
3. Do factors of health, gender and ages influence students' executive functioning (inhibitory function, working memory, and cognitive flexibility)? Researchers will compare the aerobic exercise intervention group with the no-aerobic exercise group in terms of executive function to see if and how much aerobic exercise has an effect on executive function.

Participants will:

(1) The aerobic exercise intervention group was given football and volleyball exercise intervention, and the control group was given routine school life for 3 months.

2. Record the participants before and after the intervention level of executive function.

DETAILED DESCRIPTION:
The purpose of this researchis to investigate the effects of aerobic exercise on executive function in obese children, with a focus on inhibition, working memory and cognitive flexibility. A confirmatory study was conducted to determine whether obese children have weaker executive function than normal-weight children. On the basis of existence, further studies are needed to investigate the effects of aerobic exercise on executive function in obese children.

General research objective:The aim of this study is to evaluate the effects of aerobic exercise on executive function among Obese children.Specific research objectives:1.Level:To determine the developmental level of executive function (inhibitory function, working memory, and cognitive flexibility) in normal weight and obese children aged 8-10 years.2.Effects:To investigate the effects of 12-week aerobic exercise intervention on executive function(inhibition, working memory, and cognitive flexibility) in obese children aged 8-10 years.3.Factors:To investigate whether health, gender, and age factors affect students' executive functioning (inhibition, working memory, and cognitive flexibility).

Background: 1. Childhood obesity has become one of the most urgent public health problems in the world. The obesity rate for children and adolescents aged 6 to 17 years is close to 20%. 2. Obesity not only increases the prevalence of physical diseases in children, but also has a negative impact on the development of cognitive function in this age group. 3. A function is a higher level of cognitive function, is essential for individuals to directional control behavior. It includes inhibiting function, working memory and cognitive flexibility. Cognitive developmental delays in our country the third highest number of children in the world. 4. Physical exercise on the development of cognitive function in obese children with good effect. 5. National policy guidance and the attention to Chinese children's mental health and cognitive ability. 6. Childhood is the important period of executive function development. 7. The current domestic study of obese children explore more aerobic exercise influence on obese children body composition, but the study of obesity children's executive function is not perfect. As a result, more experiments are needed to verify these conclusions.

Significance: 1. Sample selection: Obese children are a special group at a critical age. Understanding of obese children and characteristics of executive function has important value. 2. The theoretical significance: the executive function still is a hot issue in the field of psychology in the world. Research results can provide a good reference for the obese child's follow-up study. 3. Practical significance: through scientific and reasonable means to improve the quality of life in obese children and to improve the executive function, reduce the cognitive and behavioral defects. The ultimate significance is to determine whether aerobic exercise can affects the obesity children's executive function, prove the effectiveness and scientific nature of aerobic exercise.

Preliminary Results or Evidence:The conceptual framework of this study is in the theoretical framework and formed on the basis of previous research achievements, in order to solve the research questions of this study. This conceptual framework takes aerobic exercise as the independent variable and executive function as the dependent variable. Executive function includes three aspects: inhibition function, working memory function, and cognitive flexibility. Based on the theoretical basis of "Development and Practice of Physical Activity Program to Enhance Children's Executive Function" written by Chen Aiguo et al, this study investigated the effects of aerobic exercise on executive function of children aged 8 to 10 years old. This model was chosen because it was found to be very useful as a conceptual framework for predicting the effects of executive function during aerobic exercise. Therefore, it is believed that the framework model will provide a good basis for the current research.

Research Design & Methods:

Experiment 1:The levels of executive functioning among normal-weight and obese children.Executive function will be tested in obese children compared with normal-weight children. To explore the executive function of children aged 8-10 years with different body mass index (BMI). The subjects will be divided into obese group and normal weight group, and the executive function tasks of obese and normal weight children will be tested. Flanker task paradigm ,N-Back task paradigm and more-odd shifting task paradigm will be used to test the executive function, and the differences between working memory ,inhibitory control function and cognitive flexibility in different groups will be investigated. Behavioral tasks will be tested in quiet office conditions, and all three tasks will be tested using the computer program.To measure the levels of executive functioning(inhibitory function, working memory, and cognitive flexibility) in normal-weight and obese children aged 8-10 years.

experiment 2：Effects of aerobic exercise on executive function among obese children.To investigate the effects of 12-week aerobic exercise intervention on executive function (inhibitory function, working memory, and cognitive flexibility)among obese children aged 8-10 years.The participants will be divided into obese exercise group and obese control group, and the behavioral paradigm of executive function will be tested before the intervention to obtain the pre-test data. Then, the obese exercise group will be given aerobic exercise intervention for 12 weeks, and the posttest data will be collected after 12 weeks. Executive function will be tested using Flanker, N-Back and more-odd shifting task paradigms to examine the relationship between the effects of a 12-week aerobic exercise intervention on working memory , inhibitory control and Flexibility of cognition in the exercise group. The aerobic exercise intervention will be conducted in designated areas of the school playground, and the behavioral task will be tested using the computer program in quiet office conditions.

Experimental Equipment: Decathlon heart rate, height, body weight tester, equipped with E - Prime computer software Research environment: 1: aerobic exercise: Primary school playground. 2. Executive function test: Quiet computer room For the purpose of gathering data in this study, this study is delimited on the subject of the public primary schools in Jinan City. After review and discussion by expert members of the expert panel, this study determined that three computer programs that measure executive function(inhibition, working memory, and cognitive flexibility).The Intervention days regarding aerobic exercise .The present study was limited to executive function testing in children aged 8-10 years (3rd and 5th grade in Chinese primary schools) from selected primary schools where the aerobic exercise intervention was implemented and where multi-functional computer classrooms with measurable executive function were available .

ELIGIBILITY:
Inclusion Criteria:

* Age: Obese children aged 8-10 years.
* The body weight was obese or above.
* There was no history of other concomitant diseases related to obesity,Children with simple obesity.
* Normal blood pressure.
* The International Physical Activity Scale (IPAQ, Chinese version) measured participants 'physical activity in the past 7 days, with internal consistency reliability r = 0.927(Qiu NN, 2004).
* The physical condition Safety questionnaire (PAR-Q) was used to ensure that the exercise in thistest could be completed safely(Appendix2).
* Uncorrected or corrected visual acuity was normal.

Exclusion Criteria:

* In the process of the experiment, it is necessary to participate in other forms of intervention experiments. If the members of the experimental group or the control group are engaged in regular exercise or planned training, they need to be excluded from the experiment.
* If the members of the experimental group are absent from work for more than1 week, the samples will be deemed to fall off. If the members of the experimental group and the control group fail to participate in any of the data collection on time, they will be excluded.
* Before and after the experiment, the members of the experimental group or the control group who limited their movement due to sprain and other reasons were excluded.They were randomly divided into experimental group and control group.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Pre-test: executive function in normal weight children | Baseline and week 1
  Three computer programs will be used to measure executive function:1.Flanker task paradigm to measure inhibition. This test computer recorded reaction durations in milliseconds, and the test score will be calculated as the average reaction durations of the conflict and non-conflict scenarios minus.2.N-Back task paradigm to measure working memory. This test computer records the reaction time in milliseconds, and the test score is the average reaction time.3.More-odd shifting task paradigm to measure cognitive flexibility. This test computer records the reaction time in milliseconds, and the test score is the subtraction of the average reaction time of the switching condition and the non-switching condition. For each of the three tests, the computer returns Units on a Scale 0 to 1 (0= error, 1= correct) to calculate the correct rate.
Pre-test: executive function in obese children | Baseline and week 1
  Three computer programs will be used to measure executive function:1.Flanker task paradigm to measure inhibition. This test computer recorded reaction durations in milliseconds, and the test score will be calculated as the average reaction durations of the conflict and non-conflict scenarios minus.2.N-Back task paradigm to measure working memory. This test computer records the reaction time in milliseconds, and the test score is the average reaction time.3.More-odd shifting task paradigm to measure cognitive flexibility. This test computer records the reaction time in milliseconds, and the test score is the subtraction of the average reaction time of the switching condition and the non-switching condition. For each of the three tests, the computer returns Units on a Scale 0 to 1 (0= error, 1= correct) to calculate the correct rate.
After 12 weeks of executive function level of obese children | week 12
  Three computer programs will be used to measure executive function:1.Flanker task paradigm to measure inhibition. This test computer recorded reaction durations in milliseconds, and the test score will be calculated as the average reaction durations of the conflict and non-conflict scenarios minus.2.N-Back task paradigm to measure working memory. This test computer records the reaction time in milliseconds, and the test score is the average reaction time.3.More-odd shifting task paradigm to measure cognitive flexibility. This test computer records the reaction time in milliseconds, and the test score is the subtraction of the average reaction time of the switching condition and the non-switching condition. For each of the three tests, the computer returns Units on a Scale 0 to 1 (0= error, 1= correct) to calculate the correct rate.
After 12 weeks in the control group executive function level of obese children | week 12
  Three computer programs will be used to measure executive function:1.Flanker task paradigm to measure inhibition. This test computer recorded reaction durations in milliseconds, and the test score will be calculated as the average reaction durations of the conflict and non-conflict scenarios minus.2.N-Back task paradigm to measure working memory. This test computer records the reaction time in milliseconds, and the test score is the average reaction time.3.More-odd shifting task paradigm to measure cognitive flexibility. This test computer records the reaction time in milliseconds, and the test score is the subtraction of the average reaction time of the switching condition and the non-switching condition. For each of the three tests, the computer returns Units on a Scale 0 to 1 (0= error, 1= correct) to calculate the correct rate.

CONTACTS AND LOCATIONS:
Overall Officials: Borhannudin Bin Abdullah, Lecturer, Study Chair — Faculty of educational studies,,Universiti Putra Malaysia
Locations (1):
- Jinan Tangye primary School, Jinan, Shandong, China